CLINICAL TRIAL: NCT01673555
Title: A Randomized, Placebo-controlled, Study to Evaluate the Effects of GSK1278863A on Pulmonary Artery Pressure in Healthy Volunteers
Brief Title: Effects of GSK1278863A on Pulmonary Artery Pressure in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 116008
Record Dates: First submitted 2012-07-12; First posted 2012-08-28 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Anaemia
Keywords: GSK1278863; Pulmonary artery pressure
MeSH Terms: conditions — Anemia | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK1278863 5mg (Experimental): GSK1278863 5mg
  Interventions: Drug: GSK1278863
- GSK1278863 100mg (Experimental): GSK1278863 100mg
  Interventions: Drug: GSK1278863
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1278863 — GSK1278863
  Arms: GSK1278863 100mg; GSK1278863 5mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This protocol is designed to explore whether short-term therapy with GSK1278863 affects PASP under normoxic and hypoxic conditions in healthy volunteers. Healthy subjects will be evaluated using echocardiography to estimate PASP based on the velocity of the tricuspid regurgitant jet. Resting PASP will be assessed under normoxic (room air) conditions, as well as after 30 minutes' exposure to 15% O2 before, during, and after short-term treatment with GSK1278863.

DETAILED DESCRIPTION:
This is a single-center, randomized, placebo-controlled, single-blinded (subjects and investigators will be blinded, GSK internal personnel will not be blinded) study designed to test whether short-term administration (5 days) of GSK1278863 affects PASP under normoxic and hypoxic conditions in healthy volunteers. Approximately 45 healthy subjects with mild-moderate baseline tricuspid regurgitation (sufficient to allow reliable assessment of PASP) will be enrolled into this study and will provide ~15 evaluable subjects in each arm [Placebo, 5 mg, and 100 mg GSK 1278863].

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin less than and equal to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including [medical history, physical examination and laboratory tests]. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk and will not interfere with the study procedures.
* A hemoglobin value at screening between 13.5- 16 g/dL.
* Male subjects between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* BMII less than and equal to 32 kg/m2
* Single QTcB or QTcF less than 450 msec
* Screening echocardiogram of at least good quality, without clinically significant abnormalities, and with mild-moderate tricuspid regurgitation sufficient for the reliable estimation of PASP, as determined by the echocardiography core laboratory or responsible cardiologist.
* Screening PASP within the normal range under normoxic conditions.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* Any history of IV drug abuse.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 14 drinks for males or greater than 7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Strong family history of malignancy.
* Subjects with sickle cell trait.
* History of pulmonary hypertension

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2012-05-15 (Actual); Primary Completion 2012-11-19 (Actual); Study Completion 2012-11-19 (Actual)

PRIMARY OUTCOMES:
Placebo-adjusted change from baseline in PASP (estimated by transthoracic echocardiography) under normoxic conditions following 5 days of GSK1278863 | Day 5

SECONDARY OUTCOMES:
Placebo-adjusted change from baseline in PASP under normoxic and hypoxic conditions 8 hours after the first dose of study treatment | Day 1
  8 hours
Placebo-adjusted change from baseline in PASP under normoxic and hypoxic conditions following 1 day of therapy | Day 1
Placebo-adjusted change from baseline in PASP under normoxic and hypoxic conditions 8 hours after the fifth dose of study treatment | Day 5
  8 hours
Placebo-adjusted change from baseline in PASP under hypoxic conditions following 5 days of GSK1278863 | Day 5
Clinical safety and tolerability data including AE reporting, ECGs, vital signs, physical exam findings and clinical laboratory values, including hematologic parameters | Day 5
  Through-out the study
Plasma pharmacokinetics (AUC, Cmax, Tmax, T1/2, etc.) of GSK1278863 and its circulating metabolites (M2, M3, M4, M5, M6 and M13) | Day 5
  Through-out the study
RV size, RV ejection fraction, severity of tricuspid regurgitation, right ventricular outflow tract acceleration time at all time points at which echocardiograms are obtained (as data permit) | Day 5
  Exploratory outcomes; through-out the study
Biomarker/PD endpoints may include EPO, endothelin-1 and hepcidin or other markers of PHD or HIF activity, as data permit | Day 5
  Exploratory outcomes; through-out the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Olson E, Demopoulos L, Haws TF, Hu E, Fang Z, Mahar KM, Qin P, Lepore J, Bauer TA, Hiatt WR. Short-term treatment with a novel HIF-prolyl hydroxylase inhibitor (GSK1278863) failed to improve measures of performance in subjects with claudication-limited peripheral artery disease. Vasc Med. 2014 Dec;19(6):473-82. doi: 10.1177/1358863X14557151. Epub 2014 Nov 6. PMID 25377872
- See also: Results for study 116008 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116008?search=study&search_terms=116008#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register